CLINICAL TRIAL: NCT01425099
Title: An Adaptive, Two Part, Two Period, Single Sequence, Drug Interaction Study Between Dolutegravir 50 mg and Prednisone in Adult Healthy Volunteers
Brief Title: Drug Interaction Study Between Dolutegravir and Prednisone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 115696
Record Dates: First submitted 2011-08-18; First posted 2011-08-29 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-10

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): In Part 1, approximately 12 healthy subjects will receive DTG 50mg q24h for 5 days in Period 1. Subjects will then be administered DTG 50mg q24h in combination with prednisone 60mg for 5 days followed by a 5 day taper (60 mg Days 1-5, 50 mg Day 6, 40 mg Day 7, 30 mg Day 8, 20 mg Day 9 and 10 mg Day 10 - total duration of 10 days) in Period 2. There will be a screening visit 30 days before the first dose and a follow-up visit 7-14 days after the last dose of drug.
  Interventions: Drug: Dolutegravir; Drug: Prednisone
- Part 2 (Experimental): If DTG Cτ is reduced by more than 50% in Part 1, Part 2 will be carried out where a second cohort of subjects will receive DTG 50mg q24h DTG for 5 days in Period 1 followed by DTG 50mg q24h in combination with prednisone 20mg for 5 days followed by a 5 day taper (20 mg Days 1-5, 10 mg Days 6 and 7, 5 mg Days 8-10 - total duration of 10 days) in Period 2. There will be a screening visit 30 days before the first dose and a follow-up visit 7-14 days after the last dose of drug.
  Interventions: Drug: Dolutegravir; Drug: Prednisone

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir is an experimental drug in the integrase inhibitor class for the treatment of HIV.
  Other Names: GSK1349572
Drug: Prednisone — Prednisone is a commonly used corticosteroid used for a variety of medical condiitons

SUMMARY:
Dolutegravir (DTG, GSK1349572 is an integrase inhibitor that is currently in Phase 3 clinical development for the treatment of human immunodeficiency virus (HIV) infection. DTG is primarily metabolized by UDP-glucuronosyltransferase (UGT1A1) with cytochrome P450 (CYP)3A4 pathway as a minor route. Corticosteroids have demonstrated induction effects on UGTs and CYP3A4. Corticosteroids are often used in HIV-infected subjects and have the potential to reduce DTG exposure due to enzyme induction when co-administered. The primary objective of this study is to determine whether concomitant prednisone administration can affect the pharmacokinetics (PK) of DTG.

The study is a two part, two period, open label study. Part 1 will evaluate the effect of a high prednisone dose on DTG PK with the potential for an additional Part 2 depending on the results from Part 1. In Part 1, approximately 12 healthy subjects will receive DTG 50mg q24h for 5 days in Period 1. Subjects will then be administered DTG 50mg q24h in combination with prednisone 60mg for 5 days followed by a 5 day taper (total duration of 10 days) in Period 2. PK data of DTG will be obtained from Part 1 and used to inform decision making on the need for Part 2. If DTG exposure is reduced by more than 50% in Part 1, Part 2 will be carried out where a second cohort of subjects will receive DTG 50mg q24h DTG for 5 days in Period 1 followed by DTG 50mg q24h in combination with prednisone 20mg for 5 days followed by a 5 day taper (total duration of 10 days) in Period 2. Safety evaluations and serial PK samples for DTG will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug. All doses of study drugs will be taken following a moderate fat meal. This study will be conducted at one center in the United States, with healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator feels that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential or of child-bearing potential and agrees to use one of the contraception methods listed in the protocol. Female subjects must agree to use contraception until the follow-up visit.
* Body weight greater than or equal to 50 kg for males and 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, lower or upper GI bleed, inflammatory bowel disease or pancreatitis should be excluded.
* History of glaucoma, psychiatric illness, diabetes or borderline diabetes (or gestational diabetes), hypertension or other disorder that may be made worse by corticosteroid administration.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure at screening visit is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG as listed in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Composite of DTG pharmacokinetic parameters on Day 5 and Day 10: AUC(0-t), Cmax, C0, Ct, Cmin, CL/F, and t½. | Up to 24 hours post dose on Days 5 and 10
  Samples will be collected at predose and 1, 2, 3, 4, 8, 12 and 24 hours post dose

SECONDARY OUTCOMES:
Safety and tolerability parameters as assessed by change from baseline in vital signs (BP and HR), number of subjects with adverse events and toxicity grading of clinical laboratory tests | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Derived] Song IH, Borland J, Chen S, Savina P, Peppercorn AF, Piscitelli S. Effect of prednisone on the pharmacokinetics of the integrase inhibitor dolutegravir. Antimicrob Agents Chemother. 2013 Sep;57(9):4394-7. doi: 10.1128/AAC.00728-13. Epub 2013 Jul 1. PMID 23817375